CLINICAL TRIAL: NCT04337749
Title: A Study of Efficacy of Chlorhexidine Scrub, ZnO Nanoparticles Socks and the Combination of Chlorhexidine Scrub and ZnO Nanoparticles Socks for Prevention of Pitted Keratolysis
Brief Title: Chlorhexidine Scrub, ZnO Nanoparticles Socks and the Combination for Prevention of Pitted Keratolysis
Acronym: PKprevention
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: After discussing within the team, the project has been withdrawn due to the anticipated insufficiency of sample size.
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PK_prevention
Record Dates: First submitted 2020-04-05; First posted 2020-04-08 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Foot Dermatoses
Keywords: Pitted keratolysis; Prevention; Chlorhexidine solution; Zinc oxide nanoparticles
MeSH Terms: conditions — Foot Dermatoses

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Single blind controlled trial between participants, drug preparing team, doctors, investigators, and outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Chorhexidine scrub (Active Comparator): Chorhexidine scrub was given to participants for 2 weeks
  Interventions: Drug: Chorhexidine scrub
- ZnO-NPs socks (Active Comparator): ZnO-NPs socks were given to participants for 2 weeks
  Interventions: Device: ZnO-NPs socks
- Combination of chorhexidine scrub and ZnO-NPs socks (Active Comparator): Chorhexidine scrub and ZnO-NPs socks were given to participants for 2 weeks
  Interventions: Combination Product: Combination of chorhexidine scrub and ZnO-NPs socks
- Placebo (Placebo Comparator): Placebo socks were given to participants for 2 weeks
  Interventions: Device: Placebo socks

INTERVENTIONS:
Drug: Chorhexidine scrub — Chorhexidine scrub was given to patients for 2 weeks
  Arms: Chorhexidine scrub
Device: ZnO-NPs socks — ZnO-NPs socks were given to patients for 2 weeks
  Arms: ZnO-NPs socks
Combination Product: Combination of chorhexidine scrub and ZnO-NPs socks — Combination of chorhexidine scrub and ZnO-NPs socks were given to patients for 2 weeks
  Arms: Combination of chorhexidine scrub and ZnO-NPs socks
Device: Placebo socks — Placebo socks were given to patients for 2 weeks
  Arms: Placebo

SUMMARY:
This study aimed to study the efficacy of chlorhexidine scrub, zinc oxide nanoparticles (ZnO-NPs) socks and the combination of chlorhexidine scrub and ZnO-NPs socks in prevention of pitted keratolysis.

DETAILED DESCRIPTION:
Introduction Pitted keratolysis is a common skin disease, caused by various gram-positive bacteria including Corynebacterium species, Kytococcus sedentarius, Dermophilus congolensis and Actinomyces species. These bacteria create small tunnels in the stratum corneum, causing pitted lesions at plantar areas. This condition is frequent accompanied by feet malodor and is commonly found in young male adults, especially in soldiers, miners and athletes. The reported prevalence of pitted keratolysis among naval cadets in Thailand was 38.7%. Predisposing factors related to pitted keratolysis are pedal hyperhidrosis and prolonged feet occlusion. Although this condition is generally not painful, our previous study in 2018 revealed adversely affects patients' quality of life.

Regarding treatment modalities of pitted keratolysis, various medications and life-style modification have been recommended. Previous studies revealed efficacy of topical choices, including benzoyl peroxide gel, clindamycin-benzoyl peroxide gel, glycopyrrolate cream, erythromycin gel, clindamycin solution, chlorhexidine scrub and mupirocin ointment. Oral antibiotics and botulinum toxin injection were also beneficial in pitted keratolysis. As to life-style modification, wearing cotton socks and opened footwear, and proper hygiene, have also been suggested.

Zinc oxide (ZnO) has been demonstrated to exhibit antimicrobial activities against many microorganisms, such as Staphylococcus aureus, Escherichia coli, and Pseudomonas aeruginosa and fungal infections including dermatophytosis. It has been proposed that the mechanism is the generation of reactive oxygen species, such as hydrogen peroxide, on microorganism cell surfaces, thereby causing membrane dysfunction. The antimicrobial activities have been observed to vary with changes in the physical and chemical properties of ZnO, for instance, its particle size, porosity and specific surface area.

Nanobiotechnology , which is the integration of biotechnology and nanotechnology, is currently being used in drug delivery systems. The bactericidal efficacy of ZnO nanoparticles (ZnO-NPs) has been shown to improves with a decrease in their particle size. ZnO has also been shown to be is safe and compatible with human skin, which makes it a suitable additive for textiles. Research by Choopong and Sarayut established that ZnO-NP-coated socks exhibited antimicrobial activities against gram-positive (S. aureus) and gram-negative (Klebsiella pneumoniae) bacteria.

Objective This study aimed to study the efficacy of chlorhexidine scrub, zinc oxide nanoparticles (ZnO-NPs) socks and the combination of chlorhexidine scrub and ZnO-NPs socks in prevention of pitted keratolysis.

Material and Methods First-year naval rating cadets, who did not have pitted keratolysis were invited to enroll in this study. The cadets who previously received any topical treatment including topical antibiotic, antiperspirant or aluminum chloride within 6 months prior to the study were excluded. Consent was informed and obtained from all participants. Participants were assessed for behavioral risk factors and level of foot odor measured by a self-assessed visual analogue scale (VAS), using questionnaires. Clinically examination of feet was done in all subjects by treatment-blinded dermatologists. Subjects were randomly assigned either chlorhexidine scrub, ZnO-NPs socks, the combination of chlorhexidine scrub and ZnO-NPs socks, or placebo socks for 2 weeks. During the study, using of other topical treatment such as topical antibiotics, antiperspirant or aluminum chloride was not allowed. Participants who received chlorhexidine scrub were advised to wash their both soles with chlorhexidine scrub two times per day in the morning and evening. Participants who received ZnO-NPs socks or placeblo socks were asked to wear these socks everyday and at least 8 hours per day. All were able to regularly participate in physical military training during the study. Two weeks after the treatment, clinical examinations by dermatologists and the cadets' self-assessment questionnaires, including feet odor by using VAS, treatment satisfaction and adverse effects, were used to evaluate the effectiveness. Pitted lesions improvement at plantar areas, evaluated by dermatologists, was divided into no improvement, slight improvement (decrease of pitted lesions at feet for 1 level) and much improvement (decrease of pitted lesions at feet for at least 2 level). Data were analyzed using SPSS version 18 (SPSS, Inc., Chicago, IL, USA).

Duration of study: 6 months Study design: Randomized control trial

ELIGIBILITY:
Inclusion Criteria:

* First-year naval rating cadets, who did not have pitted keratolysis

Exclusion Criteria:

* The cadets who previously received any topical treatment including topical antibiotic, antiperspirant or aluminum chloride within 6 months prior to the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11-05 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
The number of patients who had pitted keratolysis after treatment | 2 weeks
  Effectiveness was evaluated

SECONDARY OUTCOMES:
The percentage of patients developed any side effect such as erythema, burning | 2 weeks
  Side effects were assessed

CONTACTS AND LOCATIONS:
Overall Officials: Charussri Leeyaphan, MD, Principal Investigator — Department of Dermatology Faculty of Medicine, Siriraj Hospital Mahidol Universit
Locations (1):
- Department of Dermatology Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Result] de Almeida HL Jr, Siqueira RN, Meireles Rda S, Rampon G, de Castro LA, Silva RM. Pitted keratolysis. An Bras Dermatol. 2016 Jan-Feb;91(1):106-8. doi: 10.1590/abd1806-4841.20164096. PMID 26982791
- [Result] Makhecha M, Dass S, Singh T, Gandhi R, Yadav T, Rathod D. Pitted keratolysis - a study of various clinical manifestations. Int J Dermatol. 2017 Nov;56(11):1154-1160. doi: 10.1111/ijd.13744. Epub 2017 Sep 18. PMID 28924971
- [Result] van der Snoek EM, Ekkelenkamp MB, Suykerbuyk JC. Pitted keratolysis; physicians' treatment and their perceptions in Dutch army personnel. J Eur Acad Dermatol Venereol. 2013 Sep;27(9):1120-6. doi: 10.1111/j.1468-3083.2012.04674.x. Epub 2012 Aug 7. PMID 22882561
- [Result] Leeyaphan C, Bunyaratavej S, Taychakhoonavudh S, Kulthanachairojana N, Pattanaprichakul P, Chanyachailert P, Ongsri P, Arunkajohnsak S, Limphoka P, Kulthanan K. Cost-effectiveness analysis and safety of erythromycin 4% gel and 4% chlorhexidine scrub for pitted keratolysis treatment. J Dermatolog Treat. 2019 Sep;30(6):627-629. doi: 10.1080/09546634.2018.1543846. Epub 2018 Dec 11. PMID 30415588
- [Result] Vlahovic TC, Dunn SP, Kemp K. The use of a clindamycin 1%-benzoyl peroxide 5% topical gel in the treatment of pitted keratolysis: a novel therapy. Adv Skin Wound Care. 2009 Dec;22(12):564-6. doi: 10.1097/01.ASW.0000363468.18117.fe. No abstract available. PMID 19935134
- [Result] Bunyaratavej S, Leeyaphan C, Chanyachailert P, Pattanaprichakul P, Ongsri P, Kulthanan K. Clinical manifestations, risk factors and quality of life in patients with pitted keratolysis: a cross-sectional study in cadets. Br J Dermatol. 2018 Nov;179(5):1220-1221. doi: 10.1111/bjd.16923. Epub 2018 Sep 14. No abstract available. PMID 29951993